CLINICAL TRIAL: NCT03257384
Title: Minimizing Peri-operative Time Delays, Maximizing Operating Room Efficiency: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-029
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Operating Room Efficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Black box recording of surgery — Time delays will be recorded from the moment the patient is draped and enters the operating room to the moment they exit the operating room.

SUMMARY:
The primary objective is to prospectively identify Operating Room (OR) time delays from the time the patient who is undergoing total laparoscopic hysterectomy enters the OR to exiting the OR. This analysis will be used to identify root cause(s) leading to OR delays and define areas for improvement. The secondary objective is to identify any improvements in OR time delays and OR utilization following implementation of a standardized framework developed to increase OR efficiency.

DETAILED DESCRIPTION:
Time delays in the operating room play a role in increasing wait time length, number of cancelled cases, health care expenditure and resources. Furthermore, it inconveniences patients and families, and delays care. Minimally invasive surgery (laparoscopy) affords same-day discharge, faster recovery, and decreased morbidity. However, performing laparoscopy requires special equipment and multiple steps during set-up that can lead to time delays if not performed efficiently. Multiple factors have been identified to contribute to inefficient care delivery including: communication error, equipment failure, lack of teamwork among nursing, surgical or anesthesia teams, and duplication of tasks.

OR delays due to inefficiency can result from a chain of intraoperative events including technical factors (ie. equipment failure or case complexity) and from non-technical human factors (ie. communication errors or lack of coordinated teamwork within and between OR teams). "The intraoperative period is the period in which the surgical team may have the most influence" on efficiency. Objective measures of intraoperative OR delays and identification of their causes can lead to the development of a standardized framework that could be generalized to any surgical discipline to improve OR efficiency.

The primary objective of this study is to prospectively identify OR time delays from the time the patient enters the OR who are undergoing total laparoscopic hysterectomy (laparoscopic gynecologic procedure that involves several potential areas for inefficiency) to case completion and exiting the OR. This analysis will be used to identify root cause(s) leading to OR delays and define areas for improvement. The causes of delays can be reported back to the team members through formative performance-based feedback. The secondary objective is to identify any improvements in OR time delays and OR utilization following implementation of a standardized framework developed to increase OR efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Total laparoscopic hysterectomy cases performed by Minimally Invasive Surgery gynecologist at St. Michael's Hospital

Exclusion Criteria:

* Procedure converted to laparotomy
* Patients who desire future child bearing potential
* Procedures performed by hysteroscopy or laparotomy
* General gynecologist surgeon (i.e. non-Minimally Invasive Surgical specialist)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include: patients undergoing total laparoscopic hysterectomy, as well as the surgeons, anesthesiologists, and nurses involved in conducting the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

PRIMARY OUTCOMES:
Operative room time delays | Recording starts when patient enters operating room and ends when they exit the room
  Time delays during a total laparoscopic hysterectomy procedure will be recorded

SECONDARY OUTCOMES:
Non-technical skills and performance of operative team | From time when patient enters operating room to time when they exit the room
  Skills and team performance will be rated using the Oxford NOTECHS Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Shore, MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03257384/Prot_000.pdf